CLINICAL TRIAL: NCT00448760
Title: A Nonrandomized Phase II Study: Feasibility and Outcome of Neo Adjuvant Chemotherapy With Oxaliplatin, Fluorodeoxyuridine (FUdR), Taxotere and Leucovorin in the Treatment of Previously Untreated Advanced Esophago-Gastric Carcinoma
Brief Title: Combination Chemotherapy in Treating Patients With Previously Untreated Stage II or Stage III Esophageal Cancer That Can Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20040006; SCCC-2003151 (Other: University of Miami Sylvester Comprehensive Cancer Center); WIRB-20051464 (Other: Western Institutional Review Board)
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Results first posted 2013-02-18 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2016-12

CONDITIONS: Esophageal Cancer
Keywords: stage II esophageal cancer; stage III esophageal cancer; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus | interventions — Docetaxel; Floxuridine; Leucovorin; Oxaliplatin; Microarray Analysis; Reverse Transcriptase Polymerase Chain Reaction

ARMS (1):
- Neoadjuvant + Adjuvant Chemotherapy (Experimental)
  Interventions: Drug: Docetaxel; Drug: Floxuridine; Drug: Leucovorin; Drug: Oxaliplatin; Genetic: Microarray analysis; Genetic: reverse transcriptase-polymerase chain reaction; Procedure: Conventional surgery

INTERVENTIONS:
Drug: Docetaxel — Intravenously, 25 mg/m2, over 30 minutes, 2 cycles
  Other Names: Taxotere
Drug: Floxuridine — Intravenuosly, 110mg/kg, continuous infusion over 24 hours, 2 cycles
  Other Names: FUdR
Drug: Leucovorin — Intravenuosly, 500mg/m2, continuous infusion over 24 hours, 2 cycles
Drug: Oxaliplatin — Intravenously, 85 mg/m2, over 2 hours, 2 cycles
Genetic: Microarray analysis — Analysis of tumor for pathologic response to protocol therapy
Genetic: reverse transcriptase-polymerase chain reaction — Analysis of tumor for pathologic response to protocol therapy
Procedure: Conventional surgery — Surgical removal of tumor for correlative studies

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin, floxuridine, docetaxel, and leucovorin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Giving chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying how well combination chemotherapy works in treating patients with previously untreated stage II or stage III esophageal cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether neoadjuvant chemotherapy comprising oxaliplatin, floxuridine, docetaxel, and leucovorin calcium improves the rate of pathologic complete response in patients with previously untreated, resectable stage II or III adenocarcinoma of the esophagus.

Secondary

* Determine the progression-free and overall survival of patients treated with this regimen.
* Determine the clinical response rates (complete response and partial response) in patients treated with this regimen.
* Evaluate thymidylate synthase (TS), mRNA gene expression, TS activity, and TS and mRNA sequence, to determine the altered spots as related to drug resistance in these patients.
* Evaluate the potential for genome-wide gene expression profiling to predict response to therapy, recurrence, progression-free survival, overall survival, and drug sensitivity and resistance in these patients.
* Define the role of 5' untranslated region (5'-UTR) on translation and drug resistance in these patients.
* Evaluate, by bone marrow aspirate analysis and flow cytometry, the initial presence of cancer cells in the marrow, and clearance of these cells after treatment with this regimen.
* Evaluate the safety of this regimen in these patients.
* Assess quality of life of patients during and after treatment with this regimen.

OUTLINE: This is a nonrandomized, open-label study.

Patients receive oxaliplatin IV over 2 hours on days 1 and 15 and docetaxel IV over 30 minutes, floxuridine IV over 24 hours, and leucovorin calcium IV over 24 hours on days 1, 8, and 15. Treatment repeats every 4 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo surgery after completion of chemotherapy. Patients who achieve pathologic complete response (pCR) receive no further chemotherapy. Patients who have not achieved a pCR receive 2 courses of adjuvant chemotherapy (same regimen as the neoadjuvant chemotherapy) beginning 3 weeks after surgery.

Patients undergo blood and tissue collection periodically for correlative studies. Samples are analyzed for thymidylate synthase (TS), mRNA gene expression, TS activity, and TS and mRNA sequence by bone marrow aspirate, flow cytometry, and quantitative reverse transcriptase-polymerase chain reaction.

Quality of life will be assessed at baseline, after neoadjuvant chemotherapy, after adjuvant therapy, and at the first 3-month follow-up visit.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 34 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of adenocarcinoma of the esophagus meeting the following criteria:

  * Stage II or III disease
  * Resectable disease
  * Previously untreated disease
* No stage I (mucosal only) or stage IV (metastatic) disease

PATIENT CHARACTERISTICS:

* WBC > 3,000/mm^3
* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Creatinine ≤ 2.0 mg/dL
* Bilirubin < 2 times normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Must have central venous access
* No other malignancy within the past 5 years
* No concurrent medical or psychiatric problem that would preclude study treatment
* No contraindications to paclitaxel

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy to the esophagus
* No oral cryotherapy (e.g., ice chips) on day 1 of each course

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2004-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bach Ardalan, MD, Study Chair — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida, United States

REFERENCES:
- [Result] Solomon N, Mezentsev D, Reis I, Lima M, Rios J, Avisar E, Franceschi D, Livingstone A, Podolsky L, Ardalan B. A phase II study of neoadjuvant and adjuvant chemotherapy with 5-fluorodeoxyuridine, leucovorin, oxaliplatin and docetaxel in the treatment of previously untreated advanced esophageal adenocarcinoma. Jpn J Clin Oncol. 2011 Apr;41(4):469-76. doi: 10.1093/jjco/hyq239. Epub 2011 Jan 21. PMID 21258083

RESULTS

PARTICIPANT FLOW:
Groups:
- Neoadjuvant + Adjuvant Chemotherapy: Floxuridine : Intravenuosly, 110mg/kg, continuous infusion over 24 hours, 2 cycles
  Leucovorin : Intravenuosly, 500mg/m2, continuous infusion over 24 hours, 2 cycles
  Conventional surgery : Surgical removal of tumor for correlative studies
  reverse transcriptase-polymerase chain reaction : Analysis of tumor for pathologic response to protocol therapy
  Docetaxel : Intravenously, 25 mg/m2, over 30 minutes, 2 cycles
  Microarray analysis : Analysis of tumor for pathologic response to protocol therapy
  Oxaliplatin : Intravenously, 85 mg/m2, over 2 hours, 2 cycles
Period: Overall Study
Arm/Group | Neoadjuvant + Adjuvant Chemotherapy
Started | 29
Completed | 26
Not Completed | 3
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: 5-Fluorodeoxyuridine, Leucovorin, Oxaliplatin and Docetaxel
Arm/Group | Single Arm
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 6
Age, Continuous [Mean (Full Range); unit: years] | 62 [50 to 80]
Gender [Count of Participants; unit: Participants]
  Female | 23
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response
Description: No evidence of cellular residual cancerous cells as evidenced by tumor tissue samples taken via surgery at the end of neo-adjuvant chemotherapy.
Time Frame: 8 - 16 weeks
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Single Arm: Floxuridine : Intravenuosly, 110mg/kg, continuous infusion over 24 hours, 2 cycles
  Leucovorin : Intravenuosly, 500mg/m2, continuous infusion over 24 hours, 2 cycles
  Conventional surgery : Surgical removal of tumor for correlative studies
  reverse transcriptase-polymerase chain reaction : Analysis of tumor for pathologic response to protocol therapy
  Docetaxel : Intravenously, 25 mg/m2, over 30 minutes, 2 cycles
  Microarray analysis : Analysis of tumor for pathologic response to protocol therapy
  Oxaliplatin : Intravenously, 85 mg/m2, over 2 hours, 2 cycles
Arm/Group | Single Arm
Number analyzed (Participants) | 24
percentage of participants | 16.7 [5.9 to 34.2]

2. Secondary Outcome: Clinical Response
Description: Overall response = Complete response (CR) + Partial Response (PR). Evaluated via endoscopic ultrasounds, PET and CT scans of the chest:
  Complete Response (CR) applies to participants complete disappearance of all measurable and evaluable disease. No new lesion. No disease related symptoms. No evidence of non-evaluable disease, including tumor markers and other laboratory values.
  Partial Response (PR) applies to participants with at least 50 percent reduction in the sum of the products of bi-dimensional perpendicular diameters of all measurable lesions. No progression of evaluable disease. No new lesions.
Time Frame: 8 - 16 weeks
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Single Arm
Number analyzed (Participants) | 24
percentage of participants | 72.4 [55.7 to 85.5]

3. Secondary Outcome: Median Progression-free Survival (PFS)
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Single Arm
Number analyzed (Participants) | 26
months | 13.6 [9 to 24]

4. Secondary Outcome: Overall Survival
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Single Arm
Number analyzed (Participants) | 29
months | 21.4 [13.6 to 32.1]

ADVERSE EVENTS:
Arm/Group | Single Arm
Serious Adverse Events (participants affected / at risk) | 25/29
Other Adverse Events (participants affected / at risk) | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=29)
Grade 3 Neutropenia (Blood and lymphatic system disorders) | 8
Grade 4 Neutropenia (Blood and lymphatic system disorders) | 3
Grade 3 Febrile Neutropenia (Blood and lymphatic system disorders) | 3
Grade 3Thrombocytopenia (Blood and lymphatic system disorders) | 1
Grade 3 Fatigue (General disorders) | 9
Grade 3 Diarrhea (Gastrointestinal disorders) | 5
Grade 3 Deep Venous Thrombosis (General disorders) | 1
Grade 3 Nausea (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes